CLINICAL TRIAL: NCT05897554
Title: Intra-arterial Thrombolysis After Successful Thrombectomy for Acute Ischemic Stroke Due to Large Vessel Occlusion in the Posterior Circulation (IAT-TOP)
Brief Title: Intra-arterial Thrombolysis After Successful Thrombectomy for Acute Ischemic Stroke in the Posterior Circulation (IAT-TOP)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Xuanwu Hospital, Beijing (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IAT-TOP
Record Dates: First submitted 2023-05-18; First posted 2023-06-09 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Acute Ischemic Stroke; Arterial Thrombosis; Posterior Circulation Brain Infarction
Keywords: Intra-arterial thrombolysis; Alteplase; Large vessel occlusion; Mechanical thrombectomy; Endovascular treatment
MeSH Terms: conditions — Ischemic Stroke; Brain Infarction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Successful mechanical thrombectomy plus intra-arterial alteplase group (Experimental): For patients in the successful MT plus intra-arterial alteplase group, after successful recanalization, neurointerventionalists administered intra-arterial thrombolysis with alteplase according to protocol. The angiographic scores will be assessed after intra-arterial thrombolysis.
  Interventions: Drug: intra-arterial alteplase
- Successful mechanical thrombectomy only group (No Intervention): For patients in the successful MT only group, the choice of MT strategy will be made by the qualified neurointerventionalist, including stent retriever, aspiration and a combination technology. Patients who underwent more than 3 thrombectomy procedures were excluded from the study. Rescue therapy was performed at the discretion of the neurointerventionalist in case of the grade of stenosis at the occlusion site was presented to be more than 70% after MT.

INTERVENTIONS:
Drug: intra-arterial alteplase — For patients in the successful MT plus intra-arterial alteplase group, after successful recanalization, neurointerventionalists administered intra-arterial thrombolysis with alteplase according to protocol. The angiographic scores will be assessed immediately after intra-arterial thrombolysis.
  Other Names: Intraarterial alteplase recombinant tissue plasminogen activator (r-tPA)
  Arms: Successful mechanical thrombectomy plus intra-arterial alteplase group

SUMMARY:
The CHOICE study suggested that the use of adjunct intra-arterial alteplase after successful endovascular reperfusion in large vessel occlusion acute ischemic strokes may result in a greater likelihood of excellent neurological outcome at 90 days. However, CHOICE was a phase-2 trial and almost exclusively enrolled anterior circulation occlusions. Therefore, data on the safety and efficacy of post-endovascular reperfusion IAT in posterior circulation stroke is lacking.

In general, anterior circulation strokes are associated with a higher risk of ICH than posterior circulation strokes. Therefore, we believe it might be safer to perform post-endovascular reperfusion IAT posterior circulation stroke. Also, there are more perforator artery in the posterior circulation, IAT would be more likely to show its benefit. Therefore, we would like to explore IA rt-PA for posterior circulation stroke after successful MT in our RCT.

In this study, one interim analysis will be performed when the enrollment volume reaches 50% of the total sample size (188 cases). DSMB will determine the premature termination or continuity of research.

ELIGIBILITY:
Inclusion Criteria:

1. Symptoms and signs compatible with ischemia in the posterior circulation;
2. Basilar artery occlusion or vertebral artery occlusion without antegrade flow to the basilar artery confirmed by computed tomographic angiography (CTA)/ magnetic resonance angiography (MRA)/ digital subtraction angiography (DSA);
3. Age ≥18 years and ≤80 years;
4. Premorbid mRS ≤1;
5. National Institutes of Health Stroke Score (NIHSS) ≥6 at admission；
6. PC-ASPECTS on CT/CTA-Source Images/MRI-DWI 6-10；
7. Treated with endovascular thrombectomy (EVT) resulting in an eTICI score ≥2b50 at end of the procedure；
8. Time from symptom onset to randomization<24 hours, including wake-up stroke and unwitnessed stroke; Time of onset of symptoms is defined as "last known well" (LKW) if symptoms are not witnessed or time of estimated basilar artery occlusion (defined as the time of sudden onset of basilar artery stroke symptoms, with no consideration of any preceding minor prodromal symptoms, as adjudicated by two neurologists) if symptoms are witnessed;
9. Informed consent obtained from the patient or his/her legal representative.

Exclusion Criteria:

1. Contraindication to Intravenous Thrombolysis (except time to treatment);
2. Complete clinical recovery in the angiography suite by end of MT procedure;
3. More than 3 passes of thrombectomy device;
4. Dissection of occluded artery or intraoperative bleeding on DSA after thrombectomy;
5. Patients in sedation and intubated patients could not be included if baseline NIHSS is not obtained by a neurologist or emergency physician prior to sedation or intubation;
6. Seizures at stroke onset which would preclude obtaining a baseline NIHSS;
7. Bilateral dilated pupils;
8. Severe contrast allergy or absolute contraindication to iodinated contrast;
9. Systolic pressure >185 mmHg or diastolic pressure >110 mmHg, and cannot be controlled by antihypertensive drugs;
10. Blood glucose <50 mg/dl (2.8 mmol/L) or >400 mg/dl (22.2 mmol/L);
11. Platelet <50*10^9/L, or aPTT >40 s, or PT >15 s;
12. Known genetic or acquired bleeding diathesis, deficiency of anticoagulant factors, or oral anticoagulant drugs and INR > 1.7, or treated with direct oral anticoagulant agents in the prior 48 hours;
13. Known Severe renal Failure as defined by a serum creatinine > 3.0 mg/dl (or 265.2 μmol/l) or glomerular Filtration Rate [GFR] <30, or patient requires hemodialysis or peritoneal dialysis;
14. Patients that cannot complete 90-day follow-up (e.g. no fixed residence, overseas patients, etc.);
15. Presumed vasculitis or septic embolization;
16. Suspicion of aortic dissection;
17. The patient has neurological disease or mental disorder before onset, which affects the assessment of the condition;
18. Females who are pregnant or in lactation;
19. Participating in other clinical trials that could confound the evaluation of the study;
20. Other circumstances that the investigator considers inappropriate for participation or may pose a significant risk to patients.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 247 (Actual)
Dates: Start 2023-08-11 (Actual); Primary Completion 2025-03-27 (Actual); Study Completion 2025-03-27 (Actual)

PRIMARY OUTCOMES:
Rate of modified Rankin Scale (mRS) score of 0-2 | 90 days (±7 days) after randomization
  The mRS score range from 0 (no disability) to 6 (death)

SECONDARY OUTCOMES:
Change of eTICI | Before intra-arterial thrombolysis vs. immediately after the completion of intra-arterial thrombolysis
  Change of eTICI after intra-arterial thrombolysis
Rate of mRS score of 0-3 | 90 days (±7 days) after randomization
  The mRS score range from 0 (no disability) to 6 (death)
Proportional distribution of modified Rankin Score | 90 days (±7 days) after randomization
  The mRS score range from 0 (no disability) to 6 (death)
Improvement of the National Institutes of Health Stroke Scale (NIHSS) score | 48 hours (±12 hours) after randomization
  The NIHSS score range from 0 (no deficit) to 42 (maximum deficit)
Rate of early neurological improvement | 48 hours (±12 hours) after randomization
  The NIHSS score 0-1 or decrease ≥8 from baseline NIHSS
Improvement of the NIHSS score | 7 days (±1 days) after randomization or discharge
  The NIHSS score range from 0 (no deficit) to 42 (maximum deficit)
EQ-5D-5L | 90 days (±7 days) after randomization
  The EQ-5D 5-Levels (EQ-5D-5L) range from 5 (no problems) to 25 (extreme problems), which deceased patients have a utility of 0.
Barthel Index | 90 days (±7 days) after randomization
  The Barthel Index range from 0 (severe disability) to 100 (no disability)
All-cause mortality | 90 days (±7 days) after randomization
  Death defined as a mRS score of 6
Rate of symptomatic intracranial hemorrhage (sICH) | Within 48 hours after randomization
  The sICH was assessed based on the Heidelberg Bleeding Classification, defined as 1) ≥4 points total NIHSS at the time of diagnosis compared to immediately before worsening; 2) ≥2 point in one NIHSS category. The rationale for this is to capture new hemorrhages that produce new neurological symptoms, making them clearly symptomatic but not causing worsening in the original stroke territory; 3) Leading to intubation/hemicraniectomy/EVD placement or other major medical/surgical intervention; 4) Absence of alternative explanation for deterioration.

CONTACTS AND LOCATIONS:
Locations (1):
- Xuanwu Hospital, Capital Medical University., Beijing, China

REFERENCES:
- [Derived] Yang B, Bai X, Yi T, Wang H, Liu Y, Ma L, Liu S, Wu S, Zhang L, Peng Y, Nogueira RG, Chen W, Jiao L. Intra-arterial Alteplase Thrombolysis After Successful Thrombectomy for Acute Ischemic Stroke in the Posterior Circulation (IAT-TOP): Study protocol and rationale. Int J Stroke. 2025 Jul;20(6):750-755. doi: 10.1177/17474930251313940. Epub 2025 Jan 23. PMID 39754489